CLINICAL TRIAL: NCT00231452
Title: Age of Exposure and Immunity to Malaria in Infants
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospital Clinic of Barcelona (Other)
Collaborators: European Commission (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple
Other Study IDs: AgeMal
Record Dates: First submitted 2005-09-30; First posted 2005-10-04 (Estimated); Last update posted 2011-10-28 (Estimated); Status verified 2011-10

CONDITIONS: Malaria
Keywords: natural acquired immunity,; clinical malaria,; P. falciparum,; age,; exposure,; neonatal immunology,; infants
MeSH Terms: conditions — Malaria | interventions — fanasil, pyrimethamine drug combination; Artesunate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Late exposure group (Experimental): Participants received monthly Sulfadoxine-Pyrimethamine (SP) plus Artesunate (AS) from 2.5-4.5 months of age and monthly placebo from 5.5-9.5 months of age.
  Interventions: Drug: Sulfadoxine-pyrimethamine (SP) + Artesunate (AS)
- Early exposure group (Experimental): Participants received monthly placebo from 2.5-4.5 months of age and monthly SP+AS from 5.5-9.5 months of age.
  Interventions: Drug: Sulfadoxine-pyrimethamine (SP) + Artesunate (AS)
- Control group (Placebo Comparator): Participants received monthly placebo from 2.5 to 9.5 months of age.
  Interventions: Drug: Sulfadoxine-pyrimethamine (SP) + Artesunate (AS)

INTERVENTIONS:
Drug: Sulfadoxine-pyrimethamine (SP) + Artesunate (AS) — Monthly chemoprophylaxis with SP (Fansidar® 500/25 mg) plus Artesunate (AS, Arsumax® 50 mg) or placebo (provided by Roche and Sanofi-Aventis) was administered according to the following age-based dosing schedule: ½ tablet of SP or placebo and ½ tablet of AS or placebo on the first day and ½ tablet of AS or placebo on the second and third days.

SUMMARY:
The overall objective is to evaluate the effect of exposure to Plasmodium (P.) falciparum erythrocytic stage antigens during different periods of infancy on the development of naturally acquired immunity (NAI).

Hypothesis: Exposure to P. falciparum prior to 5 months of age does not result in the development of NAI, while exposure to P. falciparum after 5 months of age leads to the development of NAI. The risks of clinical malaria and anaemia during the second year of life will be compared between cohorts, as well as their correlations with the type and quality of immune responses (antibodies to several P. falciparum antigens, cytokines), oxidative stress markers and host genetic factors. These results should shed light on the determinants of the development of anti-P. falciparum responses early in life and the potential constraints to early life immunisation.

ELIGIBILITY:
Inclusion Criteria:

Inclusion criteria for pregnant women:

* Healthy HIV-negative pregnant females less than 50 years of age who attend the voluntary counseling and testing (VCT) center at the Maragra or Manhiça antenatal clinic,
* Permanent residents of the Manhiça area and expecting to be living in the area with their infant for at least 2 years.

Inclusion criteria for newborn infants:

* Healthy infants, weighing >= 2 kg and having an alive mother.

Exclusion Criteria:

Exclusion criteria for pregnant women:

* Plan to leave the area in less than 2 years from the start of the study;
* Women not willing to get tested for HIV infection at the VCT center;
* Test positive for HIV;
* Not willing to provide informed consent;
* Cannot understand either Portuguese or Changana (consent forms are written in these languages).

Exclusion criteria for newborn infants:

* Any obvious congenital malformation;
* Any signs of cerebral asphyxia;
* Any obvious neonatal infection;
* Same gender Twins;
* Low birth weight (<2 kg).

Max Age: 1 Week | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 349 (Actual)
Dates: Start 2005-09; Primary Completion 2009-03 (Actual); Study Completion 2009-03 (Actual)

PRIMARY OUTCOMES:
(Clinical) Time to first or only episode of clinical malaria in the second year of life detected by passive case detection | from 12 to 24 months of age
  Global comparison between the 3 groups of the time to first or only episode of clinical malaria (according to the primary case definition) in the second year of follow up detected by passive case detection in the According-To-Protocol cohort. In addition, pairwise comparisons of the 3 groups are also presented.

SECONDARY OUTCOMES:
(Clinical) Time to first or only episode of malaria (using other case definitions), anaemia and other clinical endpoints. | 12 to 24 months of age
  Global comparison between the 3 study groups of the time to first or only episode of clinical malaria (according to the secondary case definitions) in the second year of follow up detected by passive case detection. Other endpoints include multiple episodes of malaria, time to first or only episode of anaemia, total hospital visits and prevalence of parasitaemia and anaemia at different time points. In addition, pairwise comparisons of the 3 groups are also presented.
Oxidative stress markers | multiple time points during the first two years of life (2.5, 5.5, 10.5, 15 and 24 months of age)
  Quantification of the antioxidant/pro-oxidant status over the first two years of life in relation to age of first exposure to infection.
Humoral and cellular immune responses | multiple time points during the first two years of life (2.5, 5.5, 10.5, 15 and 24 months of age)
  Quantification of antibody and cytokine responses to P. falciparum protein antigens and toxins over the first two years of life in relation to age of first exposure to infection
Host genetics | 2.5 months of age
  Analysis of haematological genetic factors, polymorphisms in genes involved in inflammatory or immunological responses to malaria and polymorphisms in genes involved in the Th1/Th2 immunological pathway.

CONTACTS AND LOCATIONS:
Overall Officials: Pedro Alonso, MD, PhD, Principal Investigator — Barcelona Center for International Health Research, Hospital Clinic/University of Barcelona; Carlota Dobaño, PhD, Principal Investigator — Barcelona Center for International Health Research, Hospital Clinic/University of Barcelona
Locations (1):
- Centro de Investigaçao em Saude da Manhiça, Manhiça, Maputo Province, Mozambique

REFERENCES:
- [Derived] Dobano C, Nhabomba AJ, Manaca MN, Berthoud T, Aguilar R, Quinto L, Barbosa A, Rodriguez MH, Jimenez A, Groves PL, Santano R, Bassat Q, Aponte JJ, Guinovart C, Doolan DL, Alonso PL. A Balanced Proinflammatory and Regulatory Cytokine Signature in Young African Children Is Associated With Lower Risk of Clinical Malaria. Clin Infect Dis. 2019 Aug 16;69(5):820-828. doi: 10.1093/cid/ciy934. PMID 30380038
- [Derived] Nhabomba AJ, Guinovart C, Jimenez A, Manaca MN, Quinto L, Cistero P, Aguilar R, Barbosa A, Rodriguez MH, Bassat Q, Aponte JJ, Mayor A, Chitnis CE, Alonso PL, Dobano C. Impact of age of first exposure to Plasmodium falciparum on antibody responses to malaria in children: a randomized, controlled trial in Mozambique. Malar J. 2014 Mar 27;13:121. doi: 10.1186/1475-2875-13-121. PMID 24674654
- [Derived] Guinovart C, Dobano C, Bassat Q, Nhabomba A, Quinto L, Manaca MN, Aguilar R, Rodriguez MH, Barbosa A, Aponte JJ, Mayor AG, Renom M, Moraleda C, Roberts DJ, Schwarzer E, Le Souef PN, Schofield L, Chitnis CE, Doolan DL, Alonso PL. The role of age and exposure to Plasmodium falciparum in the rate of acquisition of naturally acquired immunity: a randomized controlled trial. PLoS One. 2012;7(3):e32362. doi: 10.1371/journal.pone.0032362. Epub 2012 Mar 7. PMID 22412865
- See also: CISM webpage — http://www.manhica.org/
- See also: Barcelona Center for International Health Research — http://www.cresib.cat